CLINICAL TRIAL: NCT07062250
Title: Feasibility and Safety of Home Blood Count Measurement and Transfusions by Systematically Educated Patients With Acute Myeloid Leukemia
Brief Title: Feasibility and Safety of Home Blood Count Measurement and Transfusions in Patients With Acute Myeloid Leukemia
Acronym: HOME-BLOOD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Iben Husted Nielsen, Clinical nurse specialist, PhD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: p-2023-14481
Record Dates: First submitted 2025-06-05; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukaemia (AML)
Keywords: Home transfusion; Hematology; Blood transfusion; Home based treatment; Acute leukemia; Patient empowerment
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Patient Participation | interventions — Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility (Experimental): Feasibility and safety of home-based blood count measurement and transfusions
  Interventions: Device: Feasibility and safety of home-based blood count measurement and transfusions

INTERVENTIONS:
Device: Feasibility and safety of home-based blood count measurement and transfusions — Feasibility and safety of home-based blood count measurement and transfusions in patients with acute myeloid leukemia

SUMMARY:
The aim is to investigate the feasibility, safety, and complication rates of patient's self-measurement of CBC and self-administration of blood and platelet transfusions at home and examine the performance of patients conducting at-home monitoring of their blood pressure, pulse rate, saturation, and temperature before and after transfusion. Furthermore, to evaluate the health economic consequences of our innovative approach, specifically, the anticipated reduction in reliance on nurse-driven services.

This study is a single-arm feasibility study with patients newly diagnosed with Acute Myeloid Leukemia. The study will be conducted at the Department of Hematology, Rigshospitalet.

Patients are included if they are ≥ 18 years old, newly diagnosed with AML within four weeks, and scheduled to receive home-based chemotherapy. Patients are excluded if they do not speak Danish or are not assessed to be capable of performing home-based CBC measurements and administration of transfusions. Patients will be discontinued if they do not achieve remission after the second chemotherapy cycle.

Included patients will receive comprehensive training and certification to perform CBC measurements, self-administer transfusions, and monitor selected vital parameters including blood pressure, pulse rate, oxygen saturation, and temperature.

It is hypothesized that the study can demonstrate the logistic, technical, and economic feasibility and safety of educating patients with AML undergoing intensive chemotherapy, to independently conduct self-measurement of complete blood count (CBC), self-administration of transfusions at home, and examine the performance of patients conducting at-home monitoring of their blood pressure, pulse rate, saturation, and temperature before and after transfusion.

DETAILED DESCRIPTION:
Acute Myeloid Leukemia is a serious blood cancer treated with intensive chemotherapy. Around 150 patients in Denmark receive such treatment annually. Each patient undergoes 2-4 chemotherapy cycles, each followed by a 3-4 week period of bone marrow suppression, requiring frequent blood and platelet transfusions and increasing infection risk. Patients with acute myeloid leukemia, experience prolonged chemotherapy-induced pancytopenia, lasting between 2 to 4 weeks. In our existing outpatient treatment setup, patients visit the day hospital 3 times weekly for blood measurements, clinical evaluation, and transfusions with blood and platelets.

Transfusion reactions are rare, and serious complications are even less common. While some studies have explored home transfusions administered by healthcare professionals or relatives, no studies have examined self-administered home transfusions.

Patient involvement is increasingly important in cancer care. Understanding patient experiences is key to implementing safe and successful home-based care, especially in long-term, intensive treatments. Maintaining daily life and being with loved ones during treatment are highly valued by patients and families.

In this study, we aim to instruct patients to perform complete blood count measurements and self-administration of transfusions at home, thereby reducing the need for weekly visits to the hospital. However, patients will still be required to come into the hospital for blood measurements, clinical control with their responsible physician, and transfusions once weekly.

Objective To investigate the feasibility, safety, and complication rates of patients self-measurement of complete blood count and self-administration of blood and platelet transfusions at home and examine the performance of patients conducting at-home monitoring of their blood pressure, pulse rate, saturation, and temperature before and after transfusion. Furthermore, to evaluate the health economic consequences of our innovative approach, specifically, the anticipated reduction in reliance on nurse-driven services.

Design and methods This study is a single-arm feasibility study with patients newly diagnosed with acute myeloid leukemia. The study will be conducted at the Department of Hematology, Rigshospitalet.

Participants Patients are included if they are ≥ 18 years old, newly diagnosed with acute myeloid leukemia within four weeks, and scheduled to receive home-based chemotherapy. Patients are excluded if they do not speak Danish or are not assessed to be capable of performing home-based complete blood count measurements and administration of transfusions. Patients will be discontinued if they do not achieve remission after the second chemotherapy cycle.

Recruitment and Procedure Patients, n= 15 will be recruited at the outpatient clinic at the Department of Hematology, Rigshospitalet.

We will develop an educational program to facilitate certification of the patients for complete blood count self-measurements and transfusion administration. The development of the educational program will adhere to the framework outlined by the Medical Research Council for the development and evaluation of complex interventions. This education will be performed shortly after obtaining informed consent at the day hospital clinic.

The patients will receive training in drawing blood from their central venous catheter into an EDTA anticoagulated tube and in how to use HemoscreenTM. Hemoglobin and platelet values will be used to determine the need for blood and platelet transfusions. The patients will then be responsible for self-administering the blood products at the hospital under supervision by health care professionals. Patients will also learn how to administer antihistamines, acetaminophen, corticosteroids, and epinephrine either orally, subcutaneously, or intravenously following guidance from healthcare professionals at the department.

Before and after the transfusions, patients will measure their own blood pressure, pulse rate, temperature, and saturation, which is the same procedure nurses perform in relation to transfusion of blood products.

At home, patients will be responsible for independently conducting complete blood count measurements, administering transfusions, and monitoring selected vital parameters before and after transfusions, fostering their active involvement and empowerment in their treatment trajectory. Nurses at the department can always be contacted for questions and guidance. Patients will be instructed to contact the nurses in the day hospital clinic in the daytime, and the hematological ward in the evening and at night. Complete blood counts will be measured on the Hemoscreen instrument, which will feature a digital interface that allows the transfer of test results to the patient's electronic medical record at the hospital.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* newly diagnosed with AML within four weeks
* scheduled to receive home-based chemotherapy.

Exclusion Criteria:

* Patients who do not understand or speak Danish
* Incapable of performing home-based CBC measurements and administration of transfusions.
* Patients will be discontinued if they do not achieve remission after the second chemotherapy cycle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Technical Performance of the Hemoscreen Instrument | Assessed throughout each participant's enrollment period, up to 12 weeks.
  Number and classification of technical issues encountered by patients using the Hemoscreen instrument, including device malfunctions, failures, and errors in transmission of complete blood count (CBC) measurements. Recorded per transfusion event through hospital records and patient reports; categorized by issue type (e.g., hardware failure, data transmission error).
Self-Administered Blood Measurements at Home | Recorded continuously during each participant's enrollment, up to 12 weeks.
  Number of CBC measurements performed by patients at home using the Hemoscreen instrument. Extracted from hospital records and participants' self-reporting.
Self-Administered Blood and Platelet Transfusions at Home | Recorded continuously during each participant's enrollment, up to 12 weeks.
  Number of blood and platelet transfusions self-administered at home without direct hospital supervision. Extracted from hospital records and participants' self-reporting.
Replacement of Scheduled Day Hospital Visits by Home Care and Self-Testing | Recorded continuously during each participant's enrollment, up to 12 weeks.
  Number of scheduled day hospital visits replaced by successful self-testing and home transfusions. Determined by comparing hospital visit records with home care study documentation.
Vital Signs Before and After Home Transfusions | Recorded at each home transfusion event during the participant's 12-week enrollment.
  Vital parameters including temperature (°C), pulse rate (beats per minute), and blood pressure (mmHg) measured immediately before and after each home transfusion.
  Measurement: Collected by participants using standardized home monitoring devices and confirmed during nursing visits.
Extra Healthcare Visits and Hospital Admissions | Recorded continuously during each participant's enrollment, up to 12 weeks.
  Number, cause, and duration (days) of unplanned extra visits to the day hospital or inpatient ward related to transfusion or device complications. Data collected from hospital records.
Transfusion Reactions and Adverse Events | Assessed continuously during and for 24 hours post-transfusion within each participant's study period, up to 12 weeks.
  Number and severity of transfusion reactions, including serious infusion reactions necessitating hospital admission.
  Documented by clinicians and participant self-reporting; hospital admissions verified through records.
Types of Transfusion Reactions | Recorded at each transfusion event during each participant's enrollment up to 12-week study period.
  Frequency and types of transfusion reactions, categorized as fever, shivering, hypotension, hypertension, hives, nausea, pain, malaise, allergic reactions, or others.
  Recorded using a standardized transfusion reaction form during clinical assessments and participant self-reports.

SECONDARY OUTCOMES:
Change in Quality of Life scores from EORTC QLQ-C30 at baseline and post-second chemotherapy | Assessed over the course of each participant's study period, approximately 12 weeks.
  Quality of Life assessed using the validated EORTC QLQ-C30 questionnaire, which evaluates multiple dimensions of QoL in cancer patients.Patients will complete the QLQ-C30 questionnaire at two time points: at study entry (baseline) and after second chemotherapy course to monitor for any QoL deterioration during participation.
  Quality of life is measured by the validated QOL-EORTC30 questionnaire at inclusion and end of study. Data will be collected via patient self-report during scheduled visits or remotely as appropriate.
Empowerment | Assessed over the course of each participant's study period, approximately 12 weeks.
  Level of patient empowerment and satisfaction as measured by the Patient Empowerment Scale (cancer), a validated questionnaire assessing patients' sense of empowerment related to their care. Patients will complete the Patient Empowerment Scale at two time points: at study entry (baseline) and after the second chemotherapy course. Data will be collected via patient self-report during scheduled visits or remotely as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Kjeldsen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No